CLINICAL TRIAL: NCT05852886
Title: Caregiver Assisted Oral Hygiene for Individuals With Disabilities: Initial Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Disability Services, New York (Other)
Collaborators: Tufts University School of Dental Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-001
Record Dates: First submitted 2023-03-27; First posted 2023-05-10 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Oral Hygiene

STUDY DESIGN:
Intervention Model Description: First-in-human-use single arm clinical study to evaluate safety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Toothbrush (Experimental): Use of experimental toothbrush for 28 days.
  Interventions: Device: Enable Oral Hygiene System (EOHS)

INTERVENTIONS:
Device: Enable Oral Hygiene System (EOHS) — The Enable Oral Hygiene System (EOHS) is a manual toothbrush comprised of a handle and shaft with multiple surfaces of synthetic bristles extending off of the shaft at one end.

SUMMARY:
The Enable Oral Hygiene System (EOHS) is a manual toothbrush comprised of a handle and shaft with multiple surfaces of synthetic bristles extending off of the shaft at one end. EOHS is intended for a caregiver to use to remove adherent plaque and food debris from the teeth of a consumer to reduce tooth decay. Caregiver Assisted Oral Hygiene for Individuals With Disabilities: Initial Safety is a first-in-human-use single arm clinical study to evaluate the safety of EOHS. This study has been designed to assess the safety of the device during self-brushing. The primary objective of the study is to evaluate the safety of the EOHS with able-bodied individuals during self-brushing. The primary endpoint for safety is 28 days. The primary endpoint of the study will be met if there are no device failures and no Adverse Device Effects (ADEs). Subjective assessment of cleaning using the EHOS during self-brushing will also be evaluated. A total of up to 12 subjects will be enrolled in the study.

DETAILED DESCRIPTION:
Twelve subjects will be recruited to evaluate the Enable Oral Hygiene System (EOHS) for safety. Subjects will be asked to complete demographic information and a medical history. An oral exam, including evaluation of oral cavity, soft and hard tissues, will be completed following standard of care procedures. Inclusion/exclusion criteria will be evaluated and eligibility for the study will be determined. Subjects who qualify for participation in the study will receive an EOHS toothbrush with the instructions for use accompanied within the product package. Subjects will then watch an instructional video demonstrating the use of the novel toothbrush. For 28 days, subjects will use the EOHS during normal (self) brushing twice daily. Subjects will be asked to record daily impressions of comfort, ease of use, and perceived cleanliness. At the conclusion of the study, subjects will record overall subjective impressions of comfort, ease of use, and perceived cleanliness. Any device related failures, adverse events, or safety concerns will be recorded. After 28 days, an oral exam, including evaluation of oral cavity, soft and hard tissues, will be completed following standard of care procedures. Subjects will be asked to return daily and overall impression documents as well as the EOHS.

ELIGIBILITY:
Inclusion Criteria:

* Willing to attempt brushing 2 x daily.
* Write and read English.
* 18-65 years of age.

Exclusion Criteria:

* Individuals who identify as a dentist, dental student, or a dental professional.
* Any physical limitations that might compromise normal tooth brushing technique.
* Teeth with orthodontic appliances.
* Evidence of periodontal abscess or major hard or soft tissue lesions or trauma.
* Use of anti-inflammatory medications for three or more consecutive days in the previous 28 days.
* Not willing to comply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events related to toothbrush use. | 28 days
  Incidence of adverse events related to toothbrush use.
Incidence of device failure. | 28 days
  Incidence of device failure.

SECONDARY OUTCOMES:
Perception of cleanliness following use of the experimental toothbrush based on a Likert scale. | 28 days
  Likert scale based questionnaire to assess subjective assessment of cleaning.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lowenstein, MS, DMD, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No